CLINICAL TRIAL: NCT02836054
Title: Study of Degenerescence CSF Hallmarks in Older Bipolar Patients
Acronym: BPL-1318
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 38RC13.408; 2013-A00930-45 (Other: ID RCB)
Record Dates: First submitted 2013-09-20; First posted 2016-07-18 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Bipolar Disorder; Alzheimer's Disease
Keywords: biomarkers; CSF; MRI; Alzheimer's disease; bipolar disorder; cognitive functions
MeSH Terms: conditions — Bipolar Disorder; Alzheimer Disease | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with cognitive disorders (Other): lumbar punction + brain MRI
  Interventions: Procedure: lumbar puncture (LP); Procedure: brain MRI
- Patients without cognitive disorders (Other): lumbar punction + brain MRI
  Interventions: Procedure: lumbar puncture (LP); Procedure: brain MRI

INTERVENTIONS:
Procedure: lumbar puncture (LP)
Procedure: brain MRI

SUMMARY:
Analysis of 4 CSF Alzheimer's disease biomarkers (total and phosphorylated tau protein, Aß40 and Aß1-42) and morphological brain MRI in older patients (>60 year's old) with bipolar disorder, after an evaluation of their cognitive functions.

Comparison between two groups of patients : patients with cognitive disorders and patients without cognitive disorders.

The objective is to describe and compare the profile of those biomarkers in those two populations.

DETAILED DESCRIPTION:
Describe the profile of the 4 neurodegeneration's biomarkers of Alzheimer's disease dosed in the cerebrospinal fluid (Total Tau proteins, phosphorylated, Aß40 and Aß1-42) for old subjects suffering from bipolar disorder with or without cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 60 and 80
* french-speaking, reading and writing patient
* affiliation to the French Social Security
* written informed consent obtained from the patient
* agree to undergo a lumbar puncture
* easy accessibility for the lumbar puncture
* Mini Mental State Examination (MMSE) > 20
* bipolar patients :

  * type I or II
  * state of euthymia for at least 4 weeks
  * stable psychotropic drug treatment for at least 8 weeks
  * no electroconvulsive therapy during the 6 months before inclusion
* distribution in the "with cognitive disorder" or "without cognitive disorder" group is function of the result of the neuropsychological evaluation

Non-inclusion Criteria :

* severe visual or auditory disorder
* advanced lumbar osteoarthritis
* history of severe head injury, neurological disorders, diagnosed dementia
* addiction weaned for less than 12 months
* forced hospitalization in psychiatry
* MRI contraindications
* LP contraindications

Exclusion Criteria:

- at least one of the outcome measures can't be performed :

* MRI
* LP : anticoagulation, bad accessibility

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Profile 4 neurodegeneration's biomarkers of Alzheimer's disease dosed in cerebrospinal fluid of aged subjects with bipolar disorder : Total Tau proteins, phosphorylated Tau proteins, Aß40 and Aß1-42 concentration | 3 hours 50 minutes (total of the 4 primary outcome measures described)
  The mean concentration of each biomarker is measured independently. The analysis between the 2 groups is done with the profile of the 4 biomarkers, not only between the profile of one biomarker to another.

CONTACTS AND LOCATIONS:
Overall Officials: Lora COHEN, Principal Investigator — CMRR, Pavillon de Neurologie, C.H.U. de Grenoble
Locations (1):
- University Hospital, Grenoble, Grenoble, Isère, France

REFERENCES:
- [Background] Ali SO, Denicoff KD, Altshuler LL, Hauser P, Li X, Conrad AJ, Smith-Jackson EE, Leverich GS, Post RM. Relationship between prior course of illness and neuroanatomic structures in bipolar disorder: a preliminary study. Neuropsychiatry Neuropsychol Behav Neurol. 2001 Oct-Dec;14(4):227-32. PMID 11725216
- [Background] Amieva H, Le Goff M, Millet X, Orgogozo JM, Peres K, Barberger-Gateau P, Jacqmin-Gadda H, Dartigues JF. Prodromal Alzheimer's disease: successive emergence of the clinical symptoms. Ann Neurol. 2008 Nov;64(5):492-8. doi: 10.1002/ana.21509. PMID 19067364
- [Background] Augy Jennifer, Enjeux cliniques et évolutifs des troubles bipolaires. A partir d'une étude sur l'évaluation cognitive de patients bipolaires vieillissants. Thèse d'exercice. 2010.
- [Background] Bora E, Vahip S, Gonul AS, Akdeniz F, Alkan M, Ogut M, Eryavuz A. Evidence for theory of mind deficits in euthymic patients with bipolar disorder. Acta Psychiatr Scand. 2005 Aug;112(2):110-6. doi: 10.1111/j.1600-0447.2005.00570.x. PMID 15992392
- [Background] Delaloye C, Moy G, Baudois S, de Bilbao F, Remund CD, Hofer F, Ragno Paquier C, Campos L, Weber K, Gold G, Moussa A, Meiler CC, Giannakopoulos P. Cognitive features in euthymic bipolar patients in old age. Bipolar Disord. 2009 Nov;11(7):735-43. doi: 10.1111/j.1399-5618.2009.00741.x. Epub 2009 Aug 28. PMID 19719786
- [Background] Delaloye C, Moy G, de Bilbao F, Weber K, Baudois S, Haller S, Xekardaki A, Canuto A, Giardini U, Lovblad KO, Gold G, Giannakopoulos P. Longitudinal analysis of cognitive performances and structural brain changes in late-life bipolar disorder. Int J Geriatr Psychiatry. 2011 Dec;26(12):1309-18. doi: 10.1002/gps.2683. Epub 2011 Mar 10. PMID 21394788
- [Background] Doring TM, Kubo TT, Cruz LC Jr, Juruena MF, Fainberg J, Domingues RC, Gasparetto EL. Evaluation of hippocampal volume based on MR imaging in patients with bipolar affective disorder applying manual and automatic segmentation techniques. J Magn Reson Imaging. 2011 Mar;33(3):565-72. doi: 10.1002/jmri.22473. PMID 21563239
- [Background] Ewers M, Buerger K, Teipel SJ, Scheltens P, Schroder J, Zinkowski RP, Bouwman FH, Schonknecht P, Schoonenboom NS, Andreasen N, Wallin A, DeBernardis JF, Kerkman DJ, Heindl B, Blennow K, Hampel H. Multicenter assessment of CSF-phosphorylated tau for the prediction of conversion of MCI. Neurology. 2007 Dec 11;69(24):2205-12. doi: 10.1212/01.wnl.0000286944.22262.ff. PMID 18071141
- [Background] Fagan AM, Mintun MA, Shah AR, Aldea P, Roe CM, Mach RH, Marcus D, Morris JC, Holtzman DM. Cerebrospinal fluid tau and ptau(181) increase with cortical amyloid deposition in cognitively normal individuals: implications for future clinical trials of Alzheimer's disease. EMBO Mol Med. 2009 Nov;1(8-9):371-80. doi: 10.1002/emmm.200900048. PMID 20049742
- [Background] Hindley NJ, Jobst KA, King E, Barnetson L, Smith A, Haigh AM. High acceptability and low morbidity of diagnostic lumbar puncture in elderly subjects of mixed cognitive status. Acta Neurol Scand. 1995 May;91(5):405-11. doi: 10.1111/j.1600-0404.1995.tb07029.x. PMID 7639073
- [Background] Kessing LV, Nilsson FM. Increased risk of developing dementia in patients with major affective disorders compared to patients with other medical illnesses. J Affect Disord. 2003 Feb;73(3):261-9. doi: 10.1016/s0165-0327(02)00004-6. PMID 12547295
- [Background] Kessing LV, Andersen PK. Does the risk of developing dementia increase with the number of episodes in patients with depressive disorder and in patients with bipolar disorder? J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1662-6. doi: 10.1136/jnnp.2003.031773. PMID 15548477
- [Background] Li G, Sokal I, Quinn JF, Leverenz JB, Brodey M, Schellenberg GD, Kaye JA, Raskind MA, Zhang J, Peskind ER, Montine TJ. CSF tau/Abeta42 ratio for increased risk of mild cognitive impairment: a follow-up study. Neurology. 2007 Aug 14;69(7):631-9. doi: 10.1212/01.wnl.0000267428.62582.aa. PMID 17698783
- [Background] Martino DJ, Igoa A, Marengo E, Scapola M, Ais ED, Strejilevich SA. Cognitive and motor features in elderly people with bipolar disorder. J Affect Disord. 2008 Jan;105(1-3):291-5. doi: 10.1016/j.jad.2007.05.014. Epub 2007 Jun 18. PMID 17573121
- [Background] Meeks S. Bipolar disorder in the latter half of life: symptom presentation, global functioning and age of onset. J Affect Disord. 1999 Jan-Mar;52(1-3):161-7. doi: 10.1016/s0165-0327(98)00069-x. PMID 10357029
- [Background] Menecier P, Rouaud O, Arezes C, Nasr D, Menecier-Ossia L, Charvet-Blanc A, Ploton L. [Bipolar disorders and dementia: fortuitous association or filiation? A case-report and review of the literature]. Psychol Neuropsychiatr Vieil. 2007 Mar;5(1):23-34. French. PMID 17412663
- [Background] Peskind ER, Riekse R, Quinn JF, Kaye J, Clark CM, Farlow MR, Decarli C, Chabal C, Vavrek D, Raskind MA, Galasko D. Safety and acceptability of the research lumbar puncture. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19(4):220-5. doi: 10.1097/01.wad.0000194014.43575.fd. PMID 16327349
- [Background] Peskind E, Nordberg A, Darreh-Shori T, Soininen H. Safety of lumbar puncture procedures in patients with Alzheimer's disease. Curr Alzheimer Res. 2009 Jun;6(3):290-2. doi: 10.2174/156720509788486509. PMID 19519311
- [Background] Preuss UW, Watzke S, Choi JH. Diagnostic correlates of Alzheimer dementia in a U.S. Nationwide inpatient sample. Am J Geriatr Psychiatry. 2010 Sep;18(9):821-9. doi: 10.1097/JGP.0b013e3181ca3a13. PMID 20220586
- [Background] Tapiola T, Alafuzoff I, Herukka SK, Parkkinen L, Hartikainen P, Soininen H, Pirttila T. Cerebrospinal fluid beta-amyloid 42 and tau proteins as biomarkers of Alzheimer-type pathologic changes in the brain. Arch Neurol. 2009 Mar;66(3):382-9. doi: 10.1001/archneurol.2008.596. PMID 19273758
- [Background] Thomann PA, Kaiser E, Schonknecht P, Pantel J, Essig M, Schroder J. Association of total tau and phosphorylated tau 181 protein levels in cerebrospinal fluid with cerebral atrophy in mild cognitive impairment and Alzheimer disease. J Psychiatry Neurosci. 2009 Mar;34(2):136-42. PMID 19270764
- [Background] Vemuri P, Wiste HJ, Weigand SD, Knopman DS, Trojanowski JQ, Shaw LM, Bernstein MA, Aisen PS, Weiner M, Petersen RC, Jack CR Jr; Alzheimer's Disease Neuroimaging Initiative. Serial MRI and CSF biomarkers in normal aging, MCI, and AD. Neurology. 2010 Jul 13;75(2):143-51. doi: 10.1212/WNL.0b013e3181e7ca82. PMID 20625167
- [Background] Wingo AP, Harvey PD, Baldessarini RJ. Neurocognitive impairment in bipolar disorder patients: functional implications. Bipolar Disord. 2009 Mar;11(2):113-25. doi: 10.1111/j.1399-5618.2009.00665.x. PMID 19267694
- [Background] Zetterberg H, Tullhog K, Hansson O, Minthon L, Londos E, Blennow K. Low incidence of post-lumbar puncture headache in 1,089 consecutive memory clinic patients. Eur Neurol. 2010;63(6):326-30. doi: 10.1159/000311703. Epub 2010 Jun 3. PMID 20516693